CLINICAL TRIAL: NCT00629005
Title: Should We Train Strength or Skill in Post-Stroke Rehabilitation?
Brief Title: Strength Training and Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B5033-W
Record Dates: First submitted 2008-02-19; First posted 2008-03-05 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Stroke
Keywords: rehabilitation; upper extremity; motor skills
MeSH Terms: conditions — Stroke | interventions — Constraint Induced Movement Therapy; Resistance Training; Range of Motion, Articular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Constraint-Induced Movement Therapy (wear a mitt on non-paretic hand for 90% of waking hours + functional task practice for 3 hours) plus 1 hour of strength training for the arms and hands 3x/week
  Interventions: Behavioral: Constraint-Induced Movement Therapy + strength training
- Arm 2 (Active Comparator): Constraint-Induced Movement Therapy (wear a mitt on non-paretic hand for 90% of waking hours + functional task practice for 3 hours) plus non-resisted arm and hand movements for 1 hour 3x/week
  Interventions: Behavioral: Constraint-Induced Movement Therapy + range of motion

INTERVENTIONS:
Behavioral: Constraint-Induced Movement Therapy + strength training — Participants wears a mitt on non-paretic hand for 90% of waking hours and completes 3 hours of functional task practice (e.g., flipping cards, putting coins in coin slot, putting cans on a shelf) plus 1 hour of resistance elastic band exercises
  Other Names: forced use, functional task practice, progressive resistive exercise
  Arms: Arm 1
Behavioral: Constraint-Induced Movement Therapy + range of motion — Participants wears a mitt on non-paretic hand for 90% of waking hours and completes 3 hours of functional task practice (e.g., flipping cards, putting coins in coin slot, putting cans on a shelf) plus 1 hour of unresisted arm movements for
  Other Names: forced use, functional task practice
  Arms: Arm 2

SUMMARY:
People with stroke experience weakness and incoordination. Studies have shown that with functional task practice, people can increase motor control and strength to a certain extent. This study will investigate whether adding progressive resistance strength training to functional task practice modeled after Constraint-Induced Movement Therapy results in greater motor function gains than functional task practice alone

DETAILED DESCRIPTION:
To date most investigations of UE rehabilitation have examined single interventions. However, combining 2 efficacious interventions may enhance effectiveness. Both functional task training and strength training are beneficial for promoting improved upper extremity function, but they have seldom been studied as a coupled therapy. The research proposed in this project will examine the effect on UE function of adding UE resistive exercises to functional task training. Secondary aims are to examine the effect of stroke severity on the response to therapy, the interrelationship between therapy-induced neural changes and movement composition and functional changes with therapy, and test for retention of UE function gains over 6 months. Individuals with chronic hemiparesis from stroke will complete baseline testing and then be randomly assigned to either the functional task + strength training group or the functional task training alone group. Each group will train 4 hours/day, 3 days/week for 4 weeks. Each will perform 3 hours of functional task training per session. The strengthening group will then complete 1 hour of UE progressive resistance exercises while the functional task training alone group will complete gravity eliminated range of motion exercises for 1 hour. All subjects will be post-tested and then complete follow-up testing 6 months later.

ELIGIBILITY:
Inclusion Criteria:

1. age 40-85;
2. a single unilateral middle cerebral artery ischemic stroke;
3. no history of drug/alcohol abuse;
4. ability to follow 3-step commands and provide informed consent;
5. no history of other neural disorder/dysfunction (including epilepsy), no serious medical illness or refractory depression;
6. at least 300 active upper extremity elevation in scapular plane (combination of flexion and abduction);
7. ability to extend the wrist 20 degrees, and two fingers and thumb 10 degrees three times in a minute;
8. permission of physician (BRRC medical director or BRRC neurologist) to participate in strength training.

Exclusion Criteria:

1. spasticity in elbow or hand (Modified Ashworth Scale > 2);
2. Motor Activity Log32 scores >3 (which would indicate relatively good use of the upper extremity);
3. ability to complete 135 degrees shoulder elevation easily with elbow straight (e.g., doesn't hold breath, movement is fluid, little to no effort tremor observed);
4. ataxia, major sensory deficits, or hemi-inattention/neglect;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-02; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Motor Assessment - UE Subscale | Immediately after the end of therapy and 6 months later

SECONDARY OUTCOMES:
Wolf Motor Function Test | Immediately after the end of therapy and 6 months later
Cortical mapping using transcranial magnetic stimulation | Immediately after the end of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E. Nadeau, MD BS BS, Principal Investigator — North Florida/South Georgia Veterans Health System
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States